CLINICAL TRIAL: NCT01383837
Title: HIV/STI Prevention for Adolescents With Substance Use Disorders in Treatment
Acronym: STYLEnS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 6183/6622
Record Dates: First submitted 2010-08-18; First posted 2011-06-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: HIV; Sexually Transmitted Diseases
Keywords: HIV/STI; Prevention; Adolescents; Substance Use Disorders; Family-based intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STYLEnS (Experimental): Multifamily Group HIV/STI Prevention intervention or Single Family Dyad (youth and a parent)
  Interventions: Behavioral: STYLEnS
- Health Promotion (Active Comparator): Health Promotion Intervention - Adolescents only
  Interventions: Behavioral: Health Promotion

INTERVENTIONS:
Behavioral: STYLEnS — Multifamily group HIV/STI Prevention Intervention or Single Family Dyad (youth and a parent)
  Arms: STYLEnS
Behavioral: Health Promotion — Health Promotion Intervention
  Arms: Health Promotion

SUMMARY:
Adolescents with substance use disorders (SUD) are at substantial risk for contracting HIV/STIs compared to their counterparts without SUD, yet few HIV/STI sexual risk reduction interventions have been developed to meet their unique needs, and none use a family-based intervention approach, which the literature recommends as the focus for intervention for youth. Current state policies neither require providers in clinics delivering substance use treatment to offer HIV/STI sexual risk reduction nor offer providers tools or training for HIV/STI prevention. There is clear public health need to develop innovative methods of service delivery and effective strategies of HIV/STI sexual risk reduction that address multiple contexts of risk (i.e. family) for this high risk population. The current proposal addresses this need by developing a provider-delivered HIV sexual risk reduction intervention to be implemented in outpatient SUD treatment that: 1) builds the clinics' capacity to help families under their care to more comfortably address the adolescent's sexuality; 2) promotes youth's safer sex practices; and 3) reduces HIV/STI sexual risk behaviors among adolescents with SUD in care.

DETAILED DESCRIPTION:
The incidence of HIV and (sexually transmitted infections) STI continues to rise in the US among youth, and rates of HIV/STI sexual risk behaviors among adolescents with substance use disorders (SUD) are significantly higher compared with their counterparts without SUD. Yet HIV/STI sexual risk reduction is not regularly implemented within adolescent SUD treatment programs. To address this urgent public health priority, the investigators propose first to develop a manualized sexual risk reduction intervention that 1) builds community clinics' capacity to help families in their care to address systematically adolescents' sexuality; 2) promotes the youths' safer sex practices; and 3) reduces HIV/STI sexual risk behaviors among adolescents with SUD in treatment. Second, the investigators propose to pilot test the manualized intervention to examine feasibility and acceptability of implementation in real-world settings and determine optimal research parameters for such settings in preparation for a randomized clinical trial (RCT). The intervention development process will use a Community Based Participatory Research model of adaptation and development that has been successfully implemented by the PI in other settings. The investigators will conduct formative work to guide adaptation of a multi-family group HIV/STI sexual risk reduction intervention that has demonstrated efficacy with youth, ages 13-18, who have non-SUD psychiatric disorders (Project STYLE: Strengthening Today's Youth Life Experience; R01 MH63008; PI: Brown). This formative work (Phase 1 - protocol 6183) will leverage the research sample of CASALEAP, an ongoing NIDA-funded, large-scale naturalistic study of the effectiveness of outpatient SUD treatment for adolescent (R01 DA019607; PI: Hogue). The resulting new manualized intervention (STYLEnS: STYLE and Substance) then will be pilot-tested (Phase 2 - protocol 6622) with a sample of male and female adolescents with SUD (n=60) in treatment in three well-established New York City mental health outpatient treatment programs which are typical of those for adolescents with SUD and in which the investigators have active partnerships. Pilot participants will be randomly assigned to either STYLEnS or an attention control intervention (Health Promotion). Participants will receive a full-day group intervention on the day of randomization (multi-family, caregivers alone and adolescents alone), return in two weeks for an individual adolescent/caregiver dyad session, and participate in a half-day booster group session three months later. The pilot test will evaluate the feasibility and acceptability of conducting an intervention in outpatient clinics treating adolescents with SUD, examine optimal factors influencing research methods, and estimate intervention parameters for a RCT. Acceptability and feasibility will be assessed using process measures following each session as well as after the intervention is completed. The investigators will assess change in sexual risk behavior outcomes from baseline to 3 months post-intervention. This study will lay the groundwork for refining the design of a RCT of the new intervention. Implementing a HIV/STI sexual risk reduction intervention in clinics providing SUD treatment represents an innovative and potentially cost-effective approach to enable typically overburdened SUD treatment providers to address the heightened HIV/STI risk in SUD youth. This proposal responds to the need to develop HIV/STI sexual risk reduction intervention services for adolescents with SUD that can be applied in and easily disseminated to clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. are in care at the pilot sites;
2. are ages 13-24 years;
3. meet criteria for (Diagnostic Statistical Manual) DSM-IV substance abuse diagnosis (patient record);
4. have a caregiver who will consent to their study participation,
5. have a parent/family member willing to enter treatment and participate in study

Exclusion Criteria:

1. have mental retardation or pervasive developmental disorder as primary diagnosis;
2. have a medical or psychiatric illness requiring hospitalization;
3. have current psychotic features, or current suicidality;
4. are not English- or Spanish-speaking

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2010-08; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Unprotected vaginal or anal sex occasions | 3-months look back

SECONDARY OUTCOMES:
Caregiver-youth communication about sex | 3-months look back
  The Parent-Adolescent Sexual Communication Scale assesses the process and content of sexual communication between parents and adolescents. Youth and parents complete separate versions.
Caregiver-youth communication about sexual risk behaviors | 5-minutes
  The Parent-Adolescent HIV Preventive Communication Skills Scale assesses the quality and process of parent-child communication; parents and adolescents are videotaped discussing a difficult topic for 5 minutes. An observational coding system is used to match the behavior and interactive changes targeted by the Family-Based component of our intervention (e.g. I-Statements, Negative Vocalizations, and Relationship Quality). Coders will be trained and inter-rater reliability will be assessed.
Feasibility of conducting the intervention | 3-months
  Determined (yes/no) if the parent and youth attended the intervention sessions
Acceptability of the intervention | 3 months
  Adolescent and caregiver will fill out a structured post-session process measure that assesses adolescent and caregiver feedback specifically regarding intervention content, materials, format, exercises, treatment motivation, personal reactions (strengths and weaknesses, relevance, interest, satisfaction, and comfort) to receiving the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Milton L Wainberg, MD, Principal Investigator — New York State Psychiatric Institute, Columbia University
Locations (1):
- St. Lukes-Roosevelt Hospital, New York, New York, United States